CLINICAL TRIAL: NCT04793815
Title: Lung Cancer Cryo-Activation as a Novel Approach to Improve Cancer Immunogenicity and Augment Immunotherapy Efficacy
Brief Title: Lung Cancer Cryo-Activation as a Novel Approach to Augment Immunotherapy Efficacy (CRYOVATE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE20.365
Record Dates: First submitted 2021-02-24; First posted 2021-03-11 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Non-small Cell Lung Cancer Metastatic; Cryotherapy Effect
Keywords: NSCLC; Cryo-activation; Anti-PD-1
MeSH Terms: interventions — pembrolizumab; spartalizumab

STUDY DESIGN:
Intervention Model Description: Cryo-activation therapy will be performed in patients with advanced NSCLC (PD-L1≥50%) prior to ICB monotherapy in order to transform 'cold' tumors into 'warm' tumors, with the intent to improve ICB efficacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cryo-activation and anti-PD-1 monotherapy combination (Experimental)
  Interventions: Procedure: Cryo-activation; Drug: Pembrolizumab

INTERVENTIONS:
Procedure: Cryo-activation — The cryo-activation procedure involves the insertion of a cryoprobe in the tumor bed with subsequent application of very low temperatures leading to cell necrosis and tumor antigens release.
  Other Names: Endoscopic cryotherapy
Drug: Pembrolizumab — Following the cryo-activation procedure, patients will sequentially be treated with pembrolizumab (anti-PD-1) monotherapy.
  Other Names: Anti-PD-1

SUMMARY:
Cryo-activation involves the insertion of a cryoprobe in the tumor bed with subsequent cell necrosis and tumor antigens release. Such technique has the potential to induce immune-specific reactions influencing cancer cells outside of the ablated region. The addition of cryo-activation to immune-checkpoint blockers (ICB) in the advanced NSCLC setting could represent a synergistic therapeutic avenue in order to potentiate treatment responses

DETAILED DESCRIPTION:
Innovative ablation techniques have gained momentum in the last decade in order to offer alternative approaches to patients not amenable to conventional surgery. Cryoablation, a procedure by which tumor cell death is induced through cycles of freezing and thawing, represents such a pioneering technique.

The procedure involves the insertion of a cryoprobe in the tumor bed with subsequent application of very low temperatures leading to cell necrosis and tumor antigens release. In the absence of significant heat-related denaturation seen in other ablative therapy techniques (microwave, radio frequency, steam, HIFU, etc.) and as intracellular content remains in circulation following cryo-activation, it is hypothesized that such technique has the potential to induce immune-specific reactions influencing cancer cells outside of the ablated region.

This phenomenon would be reminiscent of the abscopal effect, a reaction mediated by locoregional radiotherapy exposure with the potential to trigger a systemic immune response prompting metastatic disease regression. While such immune activation would in itself be insufficient to eradicate tumor cells at distant sites, the addition of immunotherapy through checkpoint inhibition in the advanced setting could represent a synergistic therapeutic avenue in order to potentiate treatment responses in patients with NSCLC.

A phase I/II clinical trial will be conducted in order to evaluate the safety and efficacy of cryo-activation therapy in patients with previously untreated advanced NSCLC amenable to anti-PD-1 monotherapy (i.e. PD-L1 ≥50%).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥18 years of age.
* Patients must have histologically or cytologically confirmed NSCLC that is advanced/metastatic or unresectable and for which no curative therapy is available.
* Patients must present PD-L1 tumor proportion score (TPS) ≥50% in order to be eligible for first-line pembrolizumab monotherapy.
* Patients may have had prior adjuvant or neoadjuvant chemotherapy for NSCLC providing completed at least 12 months prior to relapse. Patients may not have had anti-PD-1/PD-L1 agents in the adjuvant or neoadjuvant setting.
* Patients must have an ECOG performance status 0 or 1, and a minimum life expectancy of at least 12 weeks.
* Patients must have clinically and/or radiologically documented disease with at least one lesion measurable as defined by RECIST 1.1 (excluding the lesion selected for cryo-activation). All radiology studies must be performed within 21 days prior to enrollment (within 28 days if negative). The criteria for defining measurable disease are as follows:

  * CT scan (with slice thickness of 5 mm) lesion of ≥10 mm - longest diameter (≥15 mm for nodal lesions, measured in short axis)
  * Chest x-ray ≥20 mm
  * Physical exam (using calipers) ≥10 mm
* Primary and/or secondary lung lesions or proven metastatic lymph nodes must be accessible to flexible bronchoscopy, endobronchial ultrasound (EBUS) or endoscopic ultrasound (EUS).
* Patients must have disease amenable to biopsy and be willing and able to undergo tumor biopsies at baseline, at 4 weeks following anti-PD-1 initiation and at disease progression.

Exclusion Criteria:

* Patients may NOT previously have received other immunotherapy agents, including anti-PD-1/PD-L1 or anti-CTLA-4 agent.
* Patients may NOT have received or be eligible for treatment with standard targeted therapies; patients whose tumor samples have targetable alterations, such as EGFR, ALK, BRAF or ROS1 are not eligible (K-ras mutations are not excluded).
* Patients with prior history of autoimmune disorders, active hepatitis B, untreated hepatitis C or uncontrolled human immunodeficiency virus (HIV) or untreated tuberculosis and patients treated with of immunosuppressive agents within 14 days of study drug administration are NOT eligible.
* Patients being treated with systemic corticosteroids at doses that exceed 10mg/day of prednisone (or dosing equivalents)
* Patients may not be anticoagulated with any systemic anticoagulants which cannot be held for the appropriate half-life wash-out prior to the bronchoscopic procedures (Clopidogrel, Warfarin, Heparin, etc.). Aspirin is not a contraindication.
* Patients requiring supplemental oxygen therapy at home or with saturation of less than 90% on room air.
* Allergy to topical lidocaine required for local anesthesia during bronchoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Best overall response rate (BORR; change from baseline) | every 8 weeks (until disease progression or for a maximum pembrolizumab treatment duration of 2 years), every 3 months thereafter (for up to a total of 5 years)
  Proportion of patients experiencing either complete response (CR) or partial response (PR) as their best overall response.
  The best overall response represents a change on radiological (computed tomography) follow-up and is defined as the best response from start of treatment until disease progression.

SECONDARY OUTCOMES:
Incidence of treatment-related adverse events (Safety and tolerability) | every 8 weeks (until disease progression or for a maximum pembrolizumab treatment duration of 2 years), every 3 months thereafter (for up to a total of 5 years)
  Rate of complications, adverse reactions or treatment-induced toxicities according to the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Progression-free survival (PFS) | every 8 weeks (until disease progression or for a maximum pembrolizumab treatment duration of 2 years), every 3 months thereafter (for up to a total of 5 years)
  Progression-free survival (PFS) will be calculated from the date of first anti-PD-1 dose until the date of first radiologically documented disease progression (PD) or date of death from any cause, whichever comes first, assessed up to 60 months following first anti-PD-1 dose
Overall survival (OS) | every 8 weeks (until disease progression or for a maximum pembrolizumab treatment duration of 2 years), every 3 months thereafter (for up to a total of 5 years)
  Overall survival (OS) will be calculated from the date of first anti-PD-1 dose until the date of death from any cause, assessed up to 60 months following first anti-PD-1 dose

CONTACTS AND LOCATIONS:
Overall Officials: Moishe Liberman, MD PhD, Principal Investigator — CHUM
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No